CLINICAL TRIAL: NCT06219343
Title: Non-invasive Left-sided Cervical Vagus Nerve Stimulation for Atrioventricular Reentrant Tachycardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jingye Tai (Other)
Responsible Party: Sponsor-Investigator, Jingye Tai, Principal Investigator, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2023-175-03
Record Dates: First submitted 2023-12-27; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Atrioventricular Reentrant Tachycardia
Keywords: non-invasive; vagus nerve stimulation; rapid return rhythm
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcervical non-invasive vagus nerve stimulation group (Experimental): Patient will be treated with non-invasive electrical stimulation of the left vagus nerve in the neck. After routine induction of atrioventricular reentrant tachycardia prior to radiofrequency ablation, the electrode patch was placed on the patient's left cervical vagal body surface localization, i.e., between the sternocleidomastoid muscle and the trachea where the left common carotid artery pulsation could be palpated, and resuscitation was performed using non-invasive electrical stimulation.
  Interventions: Device: Non-invasive vagus nerve stimulation

INTERVENTIONS:
Device: Non-invasive vagus nerve stimulation — Patient undergoes non-invasive vagus nerve stimulation during tachycardia episodes to see if reentry is possible

SUMMARY:
The goal of this Interventional clinical trials in atrioventricular reentrant tachycardia patients. The main question it aims to answer whether non-invasive vagus nerve stimulation could be effective in restoring rhythm.

Patients will receive non-invasive vagus nerve electrical stimulation under catheter evoked and cardiac monitoring to observe their heart rhythm changes.

DETAILED DESCRIPTION:
Participants will be treated with non-invasive electrical stimulation of the left vagus nerve in the neck. After routine induction of atrioventricular reentrant tachycardia prior to radiofrequency ablation, the electrode patch was placed on the patient's left cervical vagal body surface localization, i.e., between the sternocleidomastoid muscle and the trachea where the left common carotid artery pulsation could be palpated, and resuscitation was performed using non-invasive electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. The relevant diagnostic criteria in the Guidelines for the Diagnosis and Treatment of Supraventricular Tachycardia (svt) need to be met.
2. All need to be free of psychiatric abnormalities, verbal communication disorders, and have good compliance.
3. The patients and their families gave informed consent and signed the informed consent form.

Exclusion Criteria:

1. Does not meet the relevant diagnostic criteria in the Guidelines for the Diagnosis and Treatment of Supraventricular Tachycardia (svt).
2. Mental anomalies, verbal communication disorders, poor adherence
3. Those who do not consent to participate in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Whether the tachycardia is repetitive or not | 10minutes
  Determining whether a tachycardia is reentrant on the basis of the ambulatory electrocardiogram

SECONDARY OUTCOMES:
Parameters leading to tachycardia resumption | 10minutes
  Intensity of electrical stimuli leading to tachycardia resumption

CONTACTS AND LOCATIONS:
Overall Officials: Ai-lan Chen, Study Director — The First Hospital of Guangzhou Medical University
Locations (1):
- Ai-lan Chen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No